CLINICAL TRIAL: NCT02398253
Title: Effects of Cognitive Behavioral Therapy After a Successful Weight Loss by a Comprehensive Weight Loss Plan (NovinDiet Plan) on Weight Maintenance in Healthy Obese Female Adults: a Randomized Clinical Trial
Brief Title: Effects of Cognitive Behavioral Therapy (CBT) on Weight Maintenance After Successful Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: Tehran University of Medical Sciences (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-105
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
Keywords: weight maintenance; cognitive behavior therapy; successful weight loss
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT + Hypo-energetic Diet (Experimental)
  Interventions: Behavioral: CBT + Hypo-energetic Diet
- Hypo-energetic Diet only (Experimental)
  Interventions: Behavioral: Hypo-energetic Diet only

INTERVENTIONS:
Behavioral: CBT + Hypo-energetic Diet — This group will have cognitive behavioral therapy classes + follow the hypo-energetic diet after losing at least 10% of their body weight by using a weight loss program. They will also have monthly follow-up to 6 months by fortnightly dietician visit.
  Arms: CBT + Hypo-energetic Diet
Behavioral: Hypo-energetic Diet only — This group will receive the hypo-energetic diet only after losing at least 10% of their body weight by using a weight loss program. They will also have monthly follow-up to 6 months by fortnightly dietician visit.
  Arms: Hypo-energetic Diet only

SUMMARY:
The purpose of this study is to assess the effects of CBT after a successful weight loss by a comprehensive weight loss plan on weight maintenance in obese female adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 23-30 kg/ m² who lost at least 10% of her initial weight by the diet plan.
* Must be able to have moderate exercise.
* Must be interested to keep weight loss.

Exclusion Criteria:

* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medications that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 24 Weeks

SECONDARY OUTCOMES:
Fasting plasma glucose level | 24 weeks
lipid profiles | 48 weeks
Insulin resistance(HOMA) | 24 weeks
Waist circumference | 24 Weeks
Body mass index reduction | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Farshchi, MD, PhD, Study Chair — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ameneh Madjd, Dr., Principal Investigator — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ian A Macdonald, Prof., Principal Investigator — School of Life Sciences, The University of Nottingham; Moira A Taylor, PhD, Principal Investigator — School of Life Sciences, The University of Nottingham; Reza Malekzadeh, Prof., Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences; Alireza Delavari, MD, Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences
Locations (1):
- NovinDiet Clinic, Tehran, Iran